CLINICAL TRIAL: NCT04539418
Title: Effect of Vitamin K2 Supplementation on Vascular Calcification in Hemodialysis Patients: a Controlled Randomized Trial.
Brief Title: Vitamin K2 Supplementation and Vascular Calcification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of Salta (Other)
Responsible Party: Principal Investigator, Rocío Pérez Abúd, Principal Investigator, Catholic University of Salta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCASAL-VITK
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Renal Disease
Keywords: Hemodialysis patients; Vascular calcification; Vitamin K2
MeSH Terms: conditions — Kidney Diseases; Vascular Calcification | interventions — Vitamin K 2

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind study
Who Masked: Participant, Care Provider
Masking Description: Patients are assigned to groups through computer-generated randomization. The investigator will know about the randomization and he will give the care provider the saline or vitamin K2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamn K2 Treated patients (Active Comparator): Vitamin K2 will be given to patients randomized to ARM 1 three times a week at the end of each dialysis session to prevent it being lost through the ultrafiltration membrane (in order to use the same dialysis access) intravenously to ensure its bioavailability.
  Interventions: Drug: Vitamin K 2
- Placebo Group (Placebo Comparator): Placebo will be given to patients randomized three times a week to ARM 2 at the end of each dialysis session to prevent it being lost through the ultrafiltration membrane (in order to use the same dialysis access) intravenously to ensure its bioavailability.
  Interventions: Drug: Vitamin K 2

INTERVENTIONS:
Drug: Vitamin K 2 — Patients will be monitored during the whole protocol.
  Other Names: PLACEBO GROUP

SUMMARY:
Vascular calcification is the leading cause of death in patients with end stage renal disease (ESRD) in hemodialysis. The protein matrix Gla vitamin K dependent (MGP) is a potent inhibitor of the vascular calcification. Objective: To evaluate the effect of vitamin K2 on vascular calcification in patients on hemodialysis. Materials and Methods: A prospective, randomized, double-blind study will be performed. The study subjects will be divided into a control (1000 µl of saline) or treated group (1000 µl containing 2000 µg of Vitamin K2). Vitamin K2 will be administered three times a week intravenously at the end of each dialysis session. Blood samples for biochemical determinations and vascular calcification will be assessed before and after 6 months of treatment through carotid Doppler ultrasound.

DETAILED DESCRIPTION:
This study is designed according to the ethical reference framework for biomedical research of the Declaration of Helsinki. Its design is prospective, randomized, double blind. Study subjects will be assigned either Arm 1 or control (vial with 1000 μL of saline) or Arm 2 or treated group (vial with 1000 μL containing 2000 μg of Vitamin K2). The trial protocol was approved by the ethics committee of the Catholic University of Salta and written informed consent will be made available to all patients who agree to participate and meet the inclusion criteria. Vascular calcification will be evaluated at the beginning of the study to determine the presence of vascular calcification and at the end of the study to assess changes, if any. The carotid artery examination will be performed with a GE VIVID 5 (GE Healthcare, Little Chalfont, Buckinghamshire, UK) with a 7.5 MHz linear probe. The protocol used to obtain images is consistent with the recommendations of the American Society of Echocardiography. Longitudinal images will be obtained by means of B-mode ultrasound, the maximum and the global median intima thickness (EIM) value of the common carotid artery and the presence of carotid plaques (defined as isolated and focal areas of the abnormal intima that protrude into the lumen more than 1.5 mm or at least 50% of the surrounding total mean intimate value). The EIM represents the thickness of the intima, plus the component of the mean of the vessel wall; with an automated computerized system of the equipment, on the distal wall of both common carotid arteries, 1 cm below the carotid bulb, along a 10 mm long straight arterial segment. Patients may be stratified into 3 groups according to the EIM value: EIM patients with <0.5 mm are considered disease-free; patients with IMD between 0.6-1 mm will be considered to be non-significantly affected by the disease; patients with IMD> 1 mm will be grouped as affected by significant disease (Table 1). Therefore, carotid atherosclerosis is considered in the presence of plaques or an EIM> 1 mm. 2.5.3 Table 1. Thickness of the intima plus the component of the mean in the wall of a vessel associated or not with the presence of vascular calcification.

EIM VALUE Presence or not of vascular calcification <0,5 mm Patients without vascular calcification 0,6-1 mm Patients non-significantly affected by the disease > 1 mm Patients significantly affected by the disease

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old
* A period not less than 6 months in HD
* Life expectancy ≥ 18 months
* Signed informed consent

Exclusion Criteria:

* Patients under treatment with phosphorus chelators
* Patients who do not want to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
EFFECT OF VITAMIN K2 ON VASCULAR CALCIFICATION | 6 months
  Changes in the VC (changes in the intimate thickness of carotide artery versus baseline).
CHANGES IN THE PRODUCT PHOSPHORUS CALCIUM | 6 months
  Changes in the product phosphorus calcium versus baseline
CHANGES IN PTHi SERUM LEVELS | 6 months
  Not significant changes in PTHi serum levels versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Pérez Abud, PhD, Principal Investigator — Universidad Católica de Salta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vo TM, Disthabanchong S. Are there ways to attenuate arterial calcification and improve cardiovascular outcomes in chronic kidney disease? World J Cardiol. 2014 May 26;6(5):216-26. doi: 10.4330/wjc.v6.i5.216. PMID 24944752
- [Result] Georgianos PI, Pikilidou MI, Liakopoulos V, Balaskas EV, Zebekakis PE. Arterial stiffness in end-stage renal disease-pathogenesis, clinical epidemiology, and therapeutic potentials. Hypertens Res. 2018 May;41(5):309-319. doi: 10.1038/s41440-018-0025-5. Epub 2018 Mar 12. PMID 29531291
- [Result] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Result] Brandenburg VM, Schurgers LJ, Kaesler N, Pusche K, van Gorp RH, Leftheriotis G, Reinartz S, Koos R, Kruger T. Prevention of vasculopathy by vitamin K supplementation: can we turn fiction into fact? Atherosclerosis. 2015 May;240(1):10-6. doi: 10.1016/j.atherosclerosis.2015.02.040. Epub 2015 Feb 24. PMID 25744701
- [Result] Caluwe R, Pyfferoen L, De Boeck K, De Vriese AS. The effects of vitamin K supplementation and vitamin K antagonists on progression of vascular calcification: ongoing randomized controlled trials. Clin Kidney J. 2016 Apr;9(2):273-9. doi: 10.1093/ckj/sfv146. Epub 2015 Dec 29. PMID 26985380
- [Result] Caluwe R, Vandecasteele S, Van Vlem B, Vermeer C, De Vriese AS. Vitamin K2 supplementation in haemodialysis patients: a randomized dose-finding study. Nephrol Dial Transplant. 2014 Jul;29(7):1385-90. doi: 10.1093/ndt/gft464. Epub 2013 Nov 26. PMID 24285428
- [Result] Cannata-Andia JB, Rodriguez-Garcia M, Carrillo-Lopez N, Naves-Diaz M, Diaz-Lopez B. Vascular calcifications: pathogenesis, management, and impact on clinical outcomes. J Am Soc Nephrol. 2006 Dec;17(12 Suppl 3):S267-73. doi: 10.1681/ASN.2006080925. PMID 17130273
- [Result] Cranenburg EC, Schurgers LJ, Uiterwijk HH, Beulens JW, Dalmeijer GW, Westerhuis R, Magdeleyns EJ, Herfs M, Vermeer C, Laverman GD. Vitamin K intake and status are low in hemodialysis patients. Kidney Int. 2012 Sep;82(5):605-10. doi: 10.1038/ki.2012.191. Epub 2012 May 30. PMID 22648294
- [Result] Scheiber D, Veulemans V, Horn P, Chatrou ML, Potthoff SA, Kelm M, Schurgers LJ, Westenfeld R. High-Dose Menaquinone-7 Supplementation Reduces Cardiovascular Calcification in a Murine Model of Extraosseous Calcification. Nutrients. 2015 Aug 18;7(8):6991-7011. doi: 10.3390/nu7085318. PMID 26295257
- [Result] De Vriese AS, Caluwe R, Bailleul E, De Bacquer D, Borrey D, Van Vlem B, Vandecasteele SJ, Emmerechts J. Dose-finding study of rivaroxaban in hemodialysis patients. Am J Kidney Dis. 2015 Jul;66(1):91-8. doi: 10.1053/j.ajkd.2015.01.022. Epub 2015 Mar 21. PMID 25804678
- [Result] Goodman WG, Goldin J, Kuizon BD, Yoon C, Gales B, Sider D, Wang Y, Chung J, Emerick A, Greaser L, Elashoff RM, Salusky IB. Coronary-artery calcification in young adults with end-stage renal disease who are undergoing dialysis. N Engl J Med. 2000 May 18;342(20):1478-83. doi: 10.1056/NEJM200005183422003. PMID 10816185
- [Result] Gundberg CM, Lian JB, Booth SL. Vitamin K-dependent carboxylation of osteocalcin: friend or foe? Adv Nutr. 2012 Mar 1;3(2):149-57. doi: 10.3945/an.112.001834. PMID 22516722
- [Result] Hur DJ, Raymond GV, Kahler SG, Riegert-Johnson DL, Cohen BA, Boyadjiev SA. A novel MGP mutation in a consanguineous family: review of the clinical and molecular characteristics of Keutel syndrome. Am J Med Genet A. 2005 May 15;135(1):36-40. doi: 10.1002/ajmg.a.30680. PMID 15810001
- [Result] Inoue T, Fujita T, Kishimoto H, Makino T, Nakamura T, Nakamura T, Sato T, Yamazaki K. Randomized controlled study on the prevention of osteoporotic fractures (OF study): a phase IV clinical study of 15-mg menatetrenone capsules. J Bone Miner Metab. 2009;27(1):66-75. doi: 10.1007/s00774-008-0008-8. Epub 2008 Dec 12. PMID 19082528
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Result] Jono S, Nishizawa Y, Shioi A, Morii H. Parathyroid hormone-related peptide as a local regulator of vascular calcification. Its inhibitory action on in vitro calcification by bovine vascular smooth muscle cells. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1135-42. doi: 10.1161/01.atv.17.6.1135. PMID 9194765
- [Result] Kaesler N, Magdeleyns E, Herfs M, Schettgen T, Brandenburg V, Fliser D, Vermeer C, Floege J, Schlieper G, Kruger T. Impaired vitamin K recycling in uremia is rescued by vitamin K supplementation. Kidney Int. 2014 Aug;86(2):286-93. doi: 10.1038/ki.2013.530. Epub 2014 Jan 15. PMID 24429407
- [Result] Kruger T, Floege J. Vitamin K antagonists: beyond bleeding. Semin Dial. 2014 Jan-Feb;27(1):37-41. doi: 10.1111/sdi.12175. PMID 24400802
- [Result] London GM, Guerin AP, Marchais SJ, Metivier F, Pannier B, Adda H. Arterial media calcification in end-stage renal disease: impact on all-cause and cardiovascular mortality. Nephrol Dial Transplant. 2003 Sep;18(9):1731-40. doi: 10.1093/ndt/gfg414. PMID 12937218
- [Result] Malluche HH, Monier-Faugere MC. Understanding and managing hyperphosphatemia in patients with chronic renal disease. Clin Nephrol. 1999 Nov;52(5):267-77. PMID 10584989
- [Result] Moe SM, Chen NX. Mechanisms of vascular calcification in chronic kidney disease. J Am Soc Nephrol. 2008 Feb;19(2):213-6. doi: 10.1681/ASN.2007080854. Epub 2007 Dec 19. PMID 18094365
- [Result] Szczerba E. [Summary of the article: Patel MR, Mahaffey KW, Garg J et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med, 2011; 365: 1557-1559]. Kardiol Pol. 2012;70(1):102-3. No abstract available. Polish. PMID 22267443
- [Result] Pucaj K, Rasmussen H, Moller M, Preston T. Safety and toxicological evaluation of a synthetic vitamin K2, menaquinone-7. Toxicol Mech Methods. 2011 Sep;21(7):520-32. doi: 10.3109/15376516.2011.568983. Epub 2011 Jul 25. PMID 21781006
- [Result] Rumberger JA, Brundage BH, Rader DJ, Kondos G. Electron beam computed tomographic coronary calcium scanning: a review and guidelines for use in asymptomatic persons. Mayo Clin Proc. 1999 Mar;74(3):243-52. doi: 10.4065/74.3.243. PMID 10089993
- [Result] Schoppet M, Shroff RC, Hofbauer LC, Shanahan CM. Exploring the biology of vascular calcification in chronic kidney disease: what's circulating? Kidney Int. 2008 Feb;73(4):384-90. doi: 10.1038/sj.ki.5002696. Epub 2007 Nov 28. PMID 18046319
- [Result] Schurgers LJ, Barreto DV, Barreto FC, Liabeuf S, Renard C, Magdeleyns EJ, Vermeer C, Choukroun G, Massy ZA. The circulating inactive form of matrix gla protein is a surrogate marker for vascular calcification in chronic kidney disease: a preliminary report. Clin J Am Soc Nephrol. 2010 Apr;5(4):568-75. doi: 10.2215/CJN.07081009. Epub 2010 Feb 4. PMID 20133489
- [Result] Shroff RC, McNair R, Figg N, Skepper JN, Schurgers L, Gupta A, Hiorns M, Donald AE, Deanfield J, Rees L, Shanahan CM. Dialysis accelerates medial vascular calcification in part by triggering smooth muscle cell apoptosis. Circulation. 2008 Oct 21;118(17):1748-57. doi: 10.1161/CIRCULATIONAHA.108.783738. Epub 2008 Oct 6. PMID 18838561
- [Result] Theuwissen E, Cranenburg EC, Knapen MH, Magdeleyns EJ, Teunissen KJ, Schurgers LJ, Smit E, Vermeer C. Low-dose menaquinone-7 supplementation improved extra-hepatic vitamin K status, but had no effect on thrombin generation in healthy subjects. Br J Nutr. 2012 Nov 14;108(9):1652-7. doi: 10.1017/S0007114511007185. Epub 2012 Jan 31. PMID 22289649
- [Result] Vissers LE, Dalmeijer GW, Boer JM, Monique Verschuren WM, van der Schouw YT, Beulens JW. Intake of dietary phylloquinone and menaquinones and risk of stroke. J Am Heart Assoc. 2013 Dec 10;2(6):e000455. doi: 10.1161/JAHA.113.000455. PMID 24326161
- [Result] Westenfeld R, Krueger T, Schlieper G, Cranenburg EC, Magdeleyns EJ, Heidenreich S, Holzmann S, Vermeer C, Jahnen-Dechent W, Ketteler M, Floege J, Schurgers LJ. Effect of vitamin K2 supplementation on functional vitamin K deficiency in hemodialysis patients: a randomized trial. Am J Kidney Dis. 2012 Feb;59(2):186-95. doi: 10.1053/j.ajkd.2011.10.041. Epub 2011 Dec 9. PMID 22169620
- [Result] Winkelmayer WC, Patrick AR, Liu J, Brookhart MA, Setoguchi S. The increasing prevalence of atrial fibrillation among hemodialysis patients. J Am Soc Nephrol. 2011 Feb;22(2):349-57. doi: 10.1681/ASN.2010050459. Epub 2011 Jan 13. PMID 21233416
- [Result] Zhang YT, Tang ZY. Research progress of warfarin-associated vascular calcification and its possible therapy. J Cardiovasc Pharmacol. 2014 Jan;63(1):76-82. doi: 10.1097/FJC.0000000000000008. PMID 24072176